CLINICAL TRIAL: NCT04674280
Title: Observational Study in Multiple Sclerosis Patients Treated With Autologous Hematopoietic Stem Cell Transplantation
Acronym: OMST
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: 8410-016
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: aHSCT — Autologous haematopoietic stem cell transplantation

SUMMARY:
Observational prospective , multi-center study

Primary objective : To gain further homogenous evidence for clinical efficacy of aHSCT in patients undergoing aHSCT for MS as primary indication.

Secondary objectives:

* Safety, tolerability and toxicity of aHSCT in MS
* Quality of life and long-term disability after aHSCT
* MRI outcome after aHSCT

Primary endpoint : Time to failure to maintain a NEDA status

Secondary endpoints:

* Overall survival
* Transplant related mortality
* MRI Assessment including lesions
* Treatment-related complications

  . • Quality of life through the MS QL 54 standard assessment
* Improvement of disability

Inclusion criteria:

* Diagnosis of MS according to the 2010 revision McDonald's criteria
* Availability of a detailed clinical history about MS, including progression of disability and relapse rate in the previous 2 years, previous treatments administered
* Patients aged 18yrs or over at the time of the first aHSCT

Exclusion criteria:

* Lack of one of the above criteria
* Physical, mental, or social condition which could affect the patient from returning for follow-up visits
* Patients with cognitive impairments, who are unable to provide written, informed consent prior to any testing under this protocol, including screening and baseline investigations that are considered part of routine patient care.

Recruitment: 50 patients Recruitment period: 2 years starting from the inclusion of the 1st patient Follow-up duration: 2 years

DETAILED DESCRIPTION:
Currently, a number of new prospective comparative trials have either started or are in preparation, and the EBMT guidelines recommend treatment on a clinical trial, where available. However, some MS patients receiving aHSCT will not be eligible for these trials, which are predominantly focussed on a tightly defined group of patients with highly active RRMS. In addition, access to such trials is not universal across EBMT and therefore there is a need for structured data collection.

The investigators propose here to conduct an observational cohort study that systematically gathers experience from MS patients, for whom an adequate set of data about their clinical history and their clinical situation at baseline is available; patients will be then be followed prospectively according to their local clinical center protocol. The expectation is that local clinical protocols will be in line with the current EBMT guidelines and recommendations. Therefore, the aim will be to prospectively and non-interventionally capture a complete dataset to safety, tolerability and efficacy outcomes for aHSCT in various sub-types of MS treated in accordance with the current EBMT guidelines and recommendations. Alongside ongoing clinical trials, the investigators hope this study will meaningfully inform the evidence-base and future guidelines and recommendations for good clinical practice.

1- Study design Multi-centre, non-interventional prospective study in patients diagnosed with Multiple Sclerosis, treated with aHSCT.

2 Aims and objectives of the study

1. Primary objectives

   * To evaluate the outcome of patients undergoing aHSCT for MS as primary indication.
2. Secondary objectives

   * To gain further knowledge on safety, tolerability and toxicity of aHSCT in MS
   * To gain further knowledge on the quality of life and long-term disability of patients treated with aHSCT
   * To gain further knowledge about the MRI outcome after aHSCT

     3. Study schedule The clinical assessment at enrolment and during follow-up will be carried out according to local policies, with the expectation that centres will be working in line with the EBMT Guidelines and Recommendations for MS and immune-mediated neurological diseases. However, based on common clinical practice in patients with MS on therapy, an MRI and one neurological assessment are usually carried out yearly. Baseline MRI should be carried out within 3 months before the start of the mobilization regimen, whilst neurological examination should be accomplished as baseline assessment no more than one month before the start of the treatment.

Enrolment time is 2 years from the registration of the first patient. Follow-up is anticipated for 24 months from individual start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS according to McDonald's criteria
* Availability of a detailed clinical history about MS, including progression of disability and relapse rate in the previous 2 years, treatments administered before aHSCT, and categorization of the sub-types of MS according to current EBMT guidelines

  * Highly active relapsing remitting MS failing DMTs
  * Progressive MS with active inflammatory component. In accordance with the EBMT guidelines, this category includes both secondary and primary progressive MS with active inflammatory component.
  * Aggressive (malignant) MS not previously treated with a full course of DMT
* Patients aged 18 or over at time of first aHSCT
* Signed informed consent

Exclusion Criteria:

* Lack of one of the above criteria

  * Progressive MS without active inflammatory component, as this indication is assigned 'GNR' according to EBMT guidelines, irrespective of whether it is secondary or primary progressive.
  * Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition (physical, mental, or social) that is likely to affect the patient be able to return for the scheduled follow-up visits.
  * Patients with cognitive impairments, who are unable to provide written, informed consent prior to any testing under this protocol, including screening and baseline investigations that are considered part of routine patient care.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients wiht multiple sclerosis treated with autologous heamatopoietic stem cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Time to NEDA-3 failure | 4 years
  NEDA-3 is defined as a composite endpoint including survival without relapses, disability progression and MRI activity (new or enlarging T2 lesions or Gd-enhancing lesions on MRI).

SECONDARY OUTCOMES:
Overall survival | 4 years
  Overall survival (OS), is defined as the interval between the date of aHSCT and either the last follow-up visit or the date of death from any cause.
Transplant related mortality | 4 years
  Treatment related mortality (TRM) defined as any death following transplant that cannot be attributed to progression or relapse of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Saccardi, MD, Principal Investigator — European Society for Blood and Marrow Transplantation

IPD SHARING:
Plan to Share IPD: No